CLINICAL TRIAL: NCT04261543
Title: The Effect of High Protein and Early Resistance Exercise Versus Usual Care on Muscle Mass, Strength and Quality, Clinical Outcomes, Functional Outcomes and Quality of Life in Mechanically Ventilated Critically Ill Patients
Brief Title: The Effect of High Protein and Early Resistance Exercise Versus Usual Care in Critically Ill Patients
Acronym: EFFORT-X
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Lee Zheng Yii, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MREC ID NO: 20181115-6890
Record Dates: First submitted 2020-01-31; First posted 2020-02-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness
Keywords: protein; exercise; muscle
MeSH Terms: conditions — Critical Illness; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Protein and Early Exercise (Experimental): High protein is defined as a protein prescription of ≥2.2 gram/kg body weight; Early exercise is defined as exercise by using cycle ergometry for 45 minutes per day within 24 hours of randomization
  Interventions: Other: High protein and early exercise
- Usual Care (Active Comparator): Usual care has a protein prescription of ≤1.2 gram/kg body weight and exercise prescription as per the discretion of attending clinicians
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: High protein and early exercise — High protein is defined as protein prescription of ≥2.2 gram/kg body weight and early exercise is defined as starting cycle ergometry intervention within 24 hours of randomization
  Arms: High Protein and Early Exercise
Other: Usual Care — Usual care group has protein prescription of ≤1.2 gram/kg body weight and exercise at the discretion of attending clinicians
  Arms: Usual Care

SUMMARY:
This is a 2-arm, parallel-group, randomized controlled trial that investigates the effect of combined high protein and early resistance exercise versus usual care on muscle mass, quality and strength, clinical outcomes, functional outcomes and quality of life in mechanically ventilated critically ill patients

DETAILED DESCRIPTION:
With the advancement of critical care, about 80% of ICU patients are surviving critical illness. However, ICU survivors often experience significant post-ICU morbidities including muscle weakness and impairments in physical functioning that can persist for years. We hypothesized that early intervention with two of the most basic features of critical care: nutrition (feeding high protein) together with mobility (early resistance exercise) may help to attenuate muscle loss, thereby reducing the severity of ICU-acquired weakness and its associated physical impairments. A 2-arm, parallel-group, randomized controlled trial is proposed to investigate the effect of the combined interventions. The intervention will be conducted for up to 28 days in the ICU. Outcome measurements will be conducted by a blinded assessor at baseline (within 24 hours of randomization), Day 10 post-randomization, before hospital discharge and at 6-month post-randomization. Ultrasound and bioelectrical impedance analysis will be conducted to measure muscle mass and quality. Manual muscle testing, handgrip and knee extension strength will also be measured. Physical function will be assessed by a series of test including the six minutes walk test. Telephone interview will be conducted to administer quality of life questionnaires at 6 months. These combined simple and non-invasive interventions, if proven effective, may potentially revolutionize critical care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above
2. Mechanically ventilated and expected to remain mechanically ventilated for an additional 48 hours from screening
3. High nutritional risk (at least one of the following):

   * BMI ≤ 25 or ≥ 35
   * Moderate to severe malnutrition as defined by Subjective Global Assessment (SGA)
   * Frailty (Clinical Frailty Scale ≥ 5 from proxy)
   * SARC-F (note: 'sarc-f' is the full name, not an abbreviation) questionnaire ≥ 4
   * From point of screening, projected duration of mechanical ventilation of >4 days

Exclusion Criteria:

1. >96 continuous hours of mechanical ventilation before screening
2. Expected death or withdrawal of life-sustaining treatments within 7 days from screening
3. Pregnant (Note: post-partum and lactating patients are not excluded from the trial)
4. The responsible clinician feels that the patient either needs low or high protein
5. Patient requires parenteral nutrition only and site does not have products to reach the high protein dose group.
6. Not ambulating independently prior to illness that lead to ICU admission (use of gait aid permitted)
7. Lower extremity injury or impairments that prevents them walking prior to hospital discharge (e.g. amputation, knee/hip injury)
8. Pre-existing cognitive impairment or language barrier that prohibits outcomes assessment
9. Pre-existing primary severe systemic neuromuscular disease resulting in severe weakness pre-ICU (e.g., Guillain Barre)
10. Intracranial or spinal process affecting motor function
11. Patients in hospital >5 days prior to ICU admission
12. Not expected to stay ≥4 days after enrollment
13. Neuromuscular blocker infusion (eligible once infusion discontinued if other inclusion criteria met)
14. Lower extremity injury or impairments that prevents cycling (e.g. amputation, knee/hip injury)
15. Weight ≥150 kg
16. Physician declines enrolment for Exercise

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Rectus femoris cross-sectional area (RFCSA) | Change in RFCSA between Day 1 and Day 10 of randomization
  RFCSA measured by ultrasonography
Rectus femoris cross-sectional area (RFCSA) | Change in RFCSA between Day 1 of randomization and within 72 hours before discharge from the hospital
  RFCSA measured by ultrasonography
Rectus femoris linear depth (RF LD) | Change in RF LD between Day 1 and Day 10 of randomization
  RF LD measured by ultrasonography
Rectus femoris linear depth (RF LD) | Change in RF LD between Day 1 of randomization and within 72 hours before discharge from the hospital
  RF LD measured by ultrasonography

SECONDARY OUTCOMES:
Quadriceps muscle echogenicity | Day 1 and Day 10 of randomization, and within 72 hours before discharge from the hospital
  Quadriceps muscle echogenicity measured by ultrasonography
Quadriceps muscle pennation angle | Day 1 and Day 10 of randomization, and within 72 hours before discharge from the hospital
  Quadriceps muscle pennation angle measured by ultrasonography
Quadriceps muscle fascicle length | Day 1 and Day 10 of randomization, and within 72 hours before discharge from the hospital
  Quadriceps muscle fascicle length measured by ultrasonography
Functional Status Score for the Intensive Care Unit (FSS-ICU) | Day 1 of randomization (surrogate interview), within 72 hours before discharge from the ICU and hospital (by trained physiotherapist)
  An assessment that consist of rolling, transfer from supine to sit, sitting at the edge of bed, transfer from sit to stand and walking
Short Physical Performance Batteries (SPPB) | Within 72 hours before discharge from the ICU and hospital
  An assessment that consist of balance test, gait speed test and chair stand test
Handgrip strength | Within 72 hours before discharge from the ICU and hospital
  Handgrip strength of both hands by using handgrip dynamometer
6 minutes walk test | Within 72 hours before discharge from the hospital
  To evaluate how far the subject can walk in 6 minutes time
Manual muscle testing | Within 72 hours before discharge from the hospital
  Bilateral muscle strength for shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension and ankle dorsiflexion
Knee extension strength | Within 72 hours before discharge from the hospital
  Knee extension strength measured by Handheld Dynamometer
Mortality | Percentage of Patient who died within this ICU or hospital admission, at day 60 and 6 months post-randomization
  Percentage of patient who died
Time-to-discharge alive from the hospital | Time elapsed from randomization to hospital discharge (for a maximum of 6 months from randomization)
  Time-to-discharge alive from the hospital
Length of mechanical ventilation | Total time from start to end of mechanical ventilation for a maximum of 6 months from randomization
  Duration of mechanical ventilation
Health-related Quality of life by 36-item short form survey (SF-36) | 6 months after randomization
  SF-36 is a questionnaire that will be administered by telephone interview
Health-related Quality of life by Euro Quality of Life 5 Dimension 5 level (EQ-5D-5L) | 6 months after randomization
  EQ-5D-5L is a questionnaire that will be administered by telephone interview
Katz Activities of Daily Living (ADL) | Day 1 of randomization (surrogate interview) and 6 months after randomization (telephone interview)
  Katz ADL is a questionnaire that will be administered by either surrogate or telephone interview
Lawton Instrumental Activities of Daily Living (IADL) | Day 1 of randomization (surrogate interview) and 6 months after randomization (telephone interview)
  Lawton IADL is a questionnaire that will be administered by either surrogate or telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Yii Lee, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Heyland DK, Stapleton RD, Mourtzakis M, Hough CL, Morris P, Deutz NE, Colantuoni E, Day A, Prado CM, Needham DM. Combining nutrition and exercise to optimize survival and recovery from critical illness: Conceptual and methodological issues. Clin Nutr. 2016 Oct;35(5):1196-206. doi: 10.1016/j.clnu.2015.07.003. Epub 2015 Jul 16. PMID 26212171
- [Background] Arabi YM, Casaer MP, Chapman M, Heyland DK, Ichai C, Marik PE, Martindale RG, McClave SA, Preiser JC, Reignier J, Rice TW, Van den Berghe G, van Zanten ARH, Weijs PJM. The intensive care medicine research agenda in nutrition and metabolism. Intensive Care Med. 2017 Sep;43(9):1239-1256. doi: 10.1007/s00134-017-4711-6. Epub 2017 Apr 3. PMID 28374096